CLINICAL TRIAL: NCT01114672
Title: A Randomized Prospective, Double-Blind Placebo Controlled Study of Oral Ergocalciferol in the Treatment of Pruritis in Hemodialysis Patients
Brief Title: A Study of Oral Ergocalciferol to Treat Pruritis in Hemodialysis Patients
Acronym: CRN11
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Mary Schanler, Administrative Dietitian, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10020
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Pruritis
Keywords: Pruritis in hemodialysis patients; 25-Vitamin D in chronic kidney disease
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergocalciferol (Active Comparator)
  Interventions: Drug: 50,000 Units Ergocalciferol
- oral placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50,000 Units Ergocalciferol — 50,000 Units oral ergocalciferol to be given once weekly
  Arms: Ergocalciferol
Drug: Placebo — oral placebo once weekly
  Arms: oral placebo

SUMMARY:
Pruritis (itching) is common in many people with chronic renal failure on hemodialysis. There may be many different reasons for the pruritis. Efforts to treat the problem have not been very effective.

Vitamin D levels have been found to be low in many hemodialysis patients. Since vitamin D plays an important role in the skin and is effective in treatment of certain skin conditions that involve pruritis, it may have a role in treatment of pruritis in hemodialysis patients.

The objective of the investigators study is to determine the effect of supplementation with oral vitamin D2 (ergocalciferol) on pruritis in hemodialysis patients.

DETAILED DESCRIPTION:
Vitamin D2 is a fat soluble steroid hormone precursor which must be hydroxylated in the liver and kidney respectively to make the active form 1-25-Vitamin D. This active metabolite and related analogs have been synthesized and are frequently used in the treatment of hyperparathyroidism in patients with chronic kidney disease. However the active metabolite may not be back metabolized to the precursor forms which may have functions in other organs including the skin. Supplementation of hemodialysis patients with oral vitamin D forms would provide a source of precursors for use throughout the body.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis treatment for > 3 months
2. Subjective complaint of excessive itching

Exclusion Criteria:

1. Age < 18 years
2. Failure to provide informed consent
3. Intact PTH < 70 pg/ml or > 1,000 pg/ml
4. Serum phosphorus > 7.0
5. Serum calcium (adjusted for albumin)> 11
6. Active malignancy
7. Likelihood of imminent renal transplantation
8. Current ergocalciferol treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Study Director — Department of Nephrology, Winthrop Univ Hospital; Mary Schanler, MS, RD, Principal Investigator — Winthrop University Hospital, Outpatient Dialysis
Locations (2):
- United States (2):
  - Winthop Univ Hospital Outpatient Dialysis at Bethpage, Bethpage, New York
  - Winthrop Univ Hospital Outpatient Dialysis, Mineola, New York

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264
- [Derived] Shirazian S, Schanler M, Shastry S, Dwivedi S, Kumar M, Rice K, Miyawaki N, Ghosh S, Fishbane S. The effect of ergocalciferol on uremic pruritus severity: a randomized controlled trial. J Ren Nutr. 2013 Jul;23(4):308-14. doi: 10.1053/j.jrn.2012.12.007. Epub 2013 Feb 27. PMID 23453391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients undergoing maintenance hemodialysis were recruited from two hemodialysis facilities from 8/11/2010 to 8/1/2011.
Pre-assignment Details: Three patients failed the screening process due to exclusion criteria: One patient had PTH<70 pg/mL and two patients had serum phosphorus >7.0 mg/dL.
Groups:
- Ergocalciferol: Patients in the Ergocalciferol Arm/Group received 50,000 international units of oral Ergocalciferol once a week for a study period of 12 weeks.
- Oral Placebo: Patients in the oral placebo Arm/Group received a placebo pill once a week for a period of 12 weeks.
Period: Overall Study
Arm/Group | Ergocalciferol | Oral Placebo
Started | 25 | 25
Completed | 21 | 23
Not Completed | 4 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — transplanted | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol | Oral Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 14 | 12 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 66.1 (14.7) | 66.2 (13.7) | 66.2 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Severity of Pruritis
Description: Randomized patients will fill out a survey with questions about the degree and location of their pruritis at baseline and end of study. The total score ranged from 0-21 with 21 being the most severe and zero being the absence of any of the measures of pruritis.
  Last observation was carried forward to end of study. A decrease in the Severity of Pruritis score over time indicated an improvement in the severity of pruritis.
Time Frame: Baseline and end of study (up to 12 weeks)
Population: Number randomized in each arm 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ergocalciferol | Oral Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 10.88 (5.15) | 9.76 (5.34)
  End of study | 6.64 (6.14) | 5.12 (4.24)

ADVERSE EVENTS:
Time Frame: 15 months
Description: Only serious adverse events were intended to be collected in this study
Arm/Group | Ergocalciferol | Oral Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 2/25
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol (N=25) | Oral Placebo (N=25)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient admitted to hospital with gastroparesis. Determined not to be related to study.
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Not related to study
Abdominal distension (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to study
Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Pre-existing condition
Hepatic Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to study
Death (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to study
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Not related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No